CLINICAL TRIAL: NCT05125731
Title: Evaluation of the Effect of Parental Absence on Child's Dental Anxiety and Behaviors During Dental Treatment: A Randomized Controlled Trial
Brief Title: Effect of Parental Absence on Child's Dental Anxiety and Behaviors During Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, AYŞE IŞIL CİHAN, Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2-21-738
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Dental Anxiety; Children, Only; Dental Caries
Keywords: Behaviour management; Dental fear; Parental absence
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researcher evaluating child's behavior by watching video recordings taken during dental treatment and biostatistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Parental absence (Experimental): The parent will not be present in the dental clinic during the treatment. Parents will be instructed to wait in a waiting room outside the clinic, out of sight of the child.
  Interventions: Behavioral: Parental absence
- Parental visual support (Active Comparator): The parent will watch and wait behind a transparent barrier without disrupting the interaction between the dentist and the child. This type of separation differs from the total absence of the parent because the parent is within the child's sight.
  Interventions: Behavioral: Parental visual support
- Parental presence (Active Comparator): One of the parents will accompany the child during the dental treatment. The parent is allowed to sit next to the child without disturbing the interaction between the dentist and the child.
  Interventions: Behavioral: Parental presence

INTERVENTIONS:
Behavioral: Parental absence — Parent does not accompany the child during dental treatment
  Arms: Parental absence
Behavioral: Parental visual support — The parent does not accompany the child during the dental treatment but watches behind the glass and is seen by the child.
  Arms: Parental visual support
Behavioral: Parental presence — Parent accompanies the child during dental treatment
  Arms: Parental presence

SUMMARY:
The basis of pediatric dentistry is to provide cooperation in children with various behavioral management techniques. The presence or absence of the parent during dental treatments can be used to ensure the child's compliance with the treatment.

The aim of this study is to investigate the effect of the presence or absence of the parent on the child's dental anxiety and child's behavior during dental treatment. The secondary aim is to examine the relationship between the child's dental fear and the parent's dental fear.

Healthy children between the ages of 4-7, who have no dental experience and need restorative treatment will be included in the study. Participants will be randomly assigned to one of three study groups (Group 1: Parental absence, Group 2: Parent behind a barrier and Group 3: Parental presence).

Psychometric and projective tests will be applied to assess child's and parent's dental anxiety at the beginning of the study.

At the second appointment scheduled for the operative treatment of decayed primary molar tooth, first the child will be administered topical and local anesthesia, a rubber dam will be placed on the decayed tooth, the caries will be removed with high and low speed rotary instruments and the cavity will be restored with a compomer filling.

Children's heart rates and blood oxygen saturation will be measured by a pulse oximeter during treatment in order to evaluate dental anxiety. Children will be videotaped during treatment so that their behaviour can be evaluated later by another researcher.

After treatment, psychometric and projective tests used to measure the child's dental anxiety will be re-administered.

DETAILED DESCRIPTION:
The aim of this clinical study is:

* to determine the presence or absence of the parent during the treatment in order to ensure the cooperation of the child during the dental treatment
* to investigate the relationship between the parent's dental fear and the child's dental fear

  72 healthy children aged 4-7 will be recruited from Ankara Yıldırım Beyazıt University Faculty of Dentistry, Department of Pediatric Dentistry outpatient clinic.

Participants who met the inclusion criteria and agreed to participate will be randomly allocated to Group 1 (Parental absence), Group 2 (Parent behind a barrier) or Group 3 (Parental presence).

A simple randomization method will be used with opaque sealed envelopes containing "Group 1", "Group 2" or "Group 3" prepared separately for 4 different ages (4, 5, 6 and 7) in the study. Group allocation will be performed by an independent researcher, not involved in the study.

"Venham Picture Test" and "The Dental Subscale of the Children's Fear Survey Schedule" questionnaire will be applied to the children before and after the dental treatments.

The parent's dental anxiety will be measured with "The Corah Dental Anxiety Scale" and parent's attitude will be measured with "Parental Attitude Scale".

During the dental treatments the heart rate and the blood oxygen saturation of each participant will be recorded at 30-second intervals. The mean number of these measurements will be calculated for each of the following processes.

1. Sitting in the dental chair at the beginning of the treatment
2. Administration of topical anesthesia
3. Administration of local anesthesia
4. Caries removal with high-speed rotary instrument
5. Caries removal with low-speed rotary instrument
6. Application of dental matrix
7. Placement of dental filling material
8. Restoration finishing and polishing
9. Sitting in the dental chair at the end of the treatment

Video recordings taken during dental treatment will be watched later by a dentist who is blind to the treatment groups and the child's cooperation during treatment will be recorded using the Frankl behavioral scale.

ELIGIBILITY:
Inclusion Criteria:

* No previous dental treatment experience
* No need for urgent dental treatment
* Presence of at least one interproximal carious lesion in a primary molar tooth with a lesion depth does not exceeding 1/2 of the inner dentin radiographically and without irreversible pulp pathology

Exclusion Criteria:

* Any systemic disease, physical or mental disorder
* Uncooperative child who absolutely refuses dental treatment

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in children's dental anxiety scores on Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) at the end of the dental treatment. | 1. At the first visit- immediately after being assigned to one of the three study arms; 2. At the second visit- within 30 min after dental treatment
  The CFSS-DS is a 15-item questionnaire on various aspects of dental treatment. Each item can be given five different scores ranging from "not afraid at all (1)" to "very much afraid (5)." The CFSS-DS has a total score range of 15 to 75 and a score of 38 or more has been associated with clinical dental fear.
Mean change from baseline in children's dental anxiety scores on Venham Picture Test at the end of the dental treatment. | 1. At the first visit- immediately after being assigned to one of the three study arms; 2. At the second visit- within 30 min after dental treatment
  The Venham picture test is comprised of 8 pairs of images, where each pair represents one anxious figure and one non-anxious figure. The children are asked to select the ones that reflect their emotional state best. The anxious figure gets 1 point, and the non-anxious figure gets 0 points. The final score ranges from 0 (least anxious) to 8 (most anxious).
Heart rate measurement to assess dental anxiety | during dental treatment
  Measurement will be made with a pulse oximeter
Blood oxygen saturation measurement to assess dental anxiety | during dental treatment
  Measurement will be made with a pulse oximeter
Frankl behavioral scale to measure compliance to dental treatment | during dental treatment
  Frankl behavior scale classifies child behavior into four categories (1-definitely negative 2- negative, 3- positive and 4- definitely positive) according to the child's attitude during dental treatment.
  The video recording taken during the treatment will be evaluated by another researcher. In the "parental presence group" where the parent accompanies the child, the parent will be seated outside the camera's field of view.

SECONDARY OUTCOMES:
The Corah Dental Anxiety Scale to measure the parent's dental anxiety | At the first visit- immediately after being assigned to one of the three study arms
  The Corah Dental Anxiety Scale (DAS) is a 4-item questionnaire related to various aspects of dental treatment (Anticipating visit to the dental clinic, waiting in the dentist's office for treatment, waiting in the dental chair for drilling of teeth, waiting in the dental chair for scaling the teeth).
  Each item contains 5 possible answers. Each answer has an assigned numeric value (1-5). The sum of the values assigned for each response is the result of the test and can vary from 4 to 20 points. A score less than 9 indicates low dental anxiety. A score of 9-12 points indicates moderate dental anxiety.A score of 13-14 points indicates high dental anxiety. A score of 15-20 points indicates very high dental anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse I. Orhan, Assoc. Prof., Study Chair — Ankara Yıldırım Beyazit University Faculty of Dentistry
Locations (1):
- Ankara Yıldırım Beyazıt University Faculty of Dentistry, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Gustafsson A, Broberg A, Bodin L, Berggren U, Arnrup K. Dental behaviour management problems: the role of child personal characteristics. Int J Paediatr Dent. 2010 Jul;20(4):242-53. doi: 10.1111/j.1365-263X.2010.01046.x. PMID 20536585
- [Background] Kantaputra PN, Chiewcharnvalijkit K, Wairatpanich K, Malikaew P, Aramrattana A. Children's attitudes toward behavior management techniques used by dentists. J Dent Child (Chic). 2007 Jan-Apr;74(1):4-9. PMID 18430348
- [Background] Versloot J, Veerkamp J, Hoogstraten J. Dental anxiety and psychological functioning in children: its relationship with behaviour during treatment. Eur Arch Paediatr Dent. 2008 Feb;9 Suppl 1:36-40. doi: 10.1007/BF03262654. PMID 18328247
- [Background] Klingberg G, Berggren U, Noren JG. Dental fear in an urban Swedish child population: prevalence and concomitant factors. Community Dent Health. 1994 Dec;11(4):208-14. PMID 7850639
- [Background] Corah NL, Gale EN, Illig SJ. Assessment of a dental anxiety scale. J Am Dent Assoc. 1978 Nov;97(5):816-9. doi: 10.14219/jada.archive.1978.0394. PMID 31377
- [Background] Venham LL, Gaulin-Kremer E. A self-report measure of situational anxiety for young children. Pediatr Dent. 1979 Jun;1(2):91-6. No abstract available. PMID 399677
- [Background] Cuthbert MI, Melamed BG. A screening device: children at risk for dental fears and management problems. ASDC J Dent Child. 1982 Nov-Dec;49(6):432-6. No abstract available. PMID 6960031
- [Background] Frankl SN, Shiere FR, Fogels HR. Should the parent remain with the child in the dental operatory? J Dent Child 1962; 29: 150-163.